CLINICAL TRIAL: NCT01515527
Title: Phase II Study of Cladribine Plus Low Dose Cytarabine (LDAC) Induction Followed By Consolidation With Cladribine Plus LDAC Alternating With Decitabine in Patients With Untreated Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Cladribine Plus Low Dose Cytarabine (LDAC) Alternating With Decitabine in Patients With Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndrome (MDS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0987; NCI-2012-00145 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-01-13; First posted 2012-01-24 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Leukemia
Keywords: Leukemia; Acute myeloid leukemia; AML; myelodysplastic syndrome; MDS; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride; Decitabine; Dacogen; Cladribine; Leustatin; 2-CdA
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cladribine; Cytarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cladribine + Cytarabine Alt. with Decitabine (Experimental): Induction cycle: Cladribine intravenous (IV) over approximately 1 to 2 hours, daily on days 1-5 combined with Cytarabine subcutaneous (SQ) twice daily on days 1-10. Cytarabine should be administered approximately 3-6 hours following the start of the cladribine infusion.
  Consolidation cycle: Cladribine IV over 1 to 2 hours, daily on days 1-3 combined with Cytarabine SQ twice daily on days 1-10. Cytarabine should be administered 3-6 hours following the start of the cladribine infusion.
  Alternating with: Decitabine IV over 1 to 2 hours, daily on days 1-5.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Decitabine

INTERVENTIONS:
Drug: Cladribine — Induction cycle: 5 mg/m2 by vein on days 1 - 5 for up to 2, 28 day cycles.
  Consolidation cycle: 5 mg/m2 by vein on days 1 - 3 of cycles 2, 5, 6, 9, 10, 13, 14, 17, and 18.
  Other Names: Leustatin; 2-CdA
Drug: Cytarabine — Induction cycle: 20 mg subcutaneously twice daily on days 1-10 for up to 2, 28 day cycles.
  Consolidation cycle: 20 mg subcutaneously twice daily on days 1 - 10 of cycles 2, 5, 6, 9, 10, 13, 14, 17, and 18.
  Other Names: Ara-C; Cytosar DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Decitabine — Consolidation cycle: 20 mg/m2 by vein over 1 to 2 hours on days 1-5 of cycles 3, 4, 7, 8, 11, 12, 15, and 16.
  Other Names: Dacogen

SUMMARY:
The goal of this clinical research study is to learn if cladribine given in combination with low-dose cytarabine (LDAC) and decitabine can help control the disease in patients with AML or MDS. The safety of this drug combination will also be studied.

Cladribine is designed to interfere with the cell's ability to process DNA (the genetic material of cells). It can also insert itself into the DNA of cancer cells to stop them from growing and repairing themselves.

Cytarabine is designed to insert itself into DNA of cancer cells to stop them from growing and repairing themselves.

Decitabine is designed to damage the DNA of cells, which may cause cancer cells to die.

This is an investigational study. Cladribine is FDA approved and commercially available for use in patients with hairy cell leukemia. Its use in patients with AML is investigational.

Cytarabine is FDA approved and commercially available for use in patients with AML.

Decitabine is FDA approved and commercially available for use in patients with MDS. Its use for patients with AML is investigational.

Up to 160 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are eligible to take part in this study, you will receive 1 or 2 cycles of induction therapy followed by up to 17 cycles of consolidation therapy. Each study cycle is 4 weeks.

Induction Cycles:

On Days 1-5, you will receive cladribine by vein over 1-2 hours.

On Days 1-10, you will give yourself the cytarabine by injection twice a day about 12 hours apart. You will receive instructions on how give yourself the injections.

You may receive up to 2 cycles at this dose and schedule.

Consolidation Cycles:

Consolidation cycles will begin on Cycle 2 regardless of how many cycles you received of induction therapy.

During Cycles 2, 5, 6, 9, 10, 13, 14, 17, and 18:

* On Days 1-3, you will receive cladribine by vein over 1-2 hours.
* On Days 1-10, you will give yourself cytarabine by injection twice daily starting 3 to 6 hours after the start of the cladribine infusion.

Cycles 3, 4, 7, 8, 11, 12, 15, and 16:

°On Days 1-5, you will receive decitabine by vein over 1-2 hours each day.

Length of Treatment:

You may continue taking the study drugs for up to 18 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over when you have completed follow-up.

Study Visits:

On Day 1 of every cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.

On Day 21 (+/- 7days) of the induction cycle, you may have a bone marrow aspirate to check the status of the disease. After that, you will have a bone marrow aspirate every 2 weeks (or more often if your doctor feels it is necessary). If your routine blood tests show that there is still leukemia, you may not need to have the bone marrow samples collected.

Blood (about 1-2 teaspoons) will be drawn for routine tests at least 1 time weekly until remission, then every 2-4 weeks during treatment, the every 4-8 weeks while you are on the study.

Follow-Up Visits:

When you are off treatment, every 6 -12 months you will be contacted by a member of the study staff. You will be asked about any side effects you may be having. The phone calls will take about 5-10 minutes. You will continue to be called for as long as possible.

ELIGIBILITY:
Cohort 1

Inclusion Criteria:

1. Patients with previously untreated AML or high risk MDS (>/= 10 % blasts or IPSS >/= intermediate-2). Prior therapy with hydroxyurea, hematopoietic growth factors, azacytidine, ATRA, or total dose of cytarabine up to 2g is allowed. Patients with history of MDS transformed to AML are eligible regardless of their prior therapy for MDS provided this will be their first induction therapy for AML.
2. Age >/= 60 years. Patients aged < 60 years who are unsuitable for standard induction therapy may be eligible after discussion with PI
3. Adequate organ function as defined below:

   * liver function (bilirubin < 2mg/dL, AST and/or ALT <3 x ULN)
   * kidney function (creatinine < 1.5 x ULN ).
4. ECOG performance status of ≤ 2.
5. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
6. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient is required prior to their enrollment on the protocol.
7. Prior therapy with decitabine will be allowed unless the patient experienced progression to AML while being treated with decitabine.

Exclusion Criteria:

1. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
2. Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patient with documented hypersensitivity to any of the components of the chemotherapy program.
4. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.

Cohort 2

Inclusion Criteria:

8. Patients with previously untreated AML who are not currently eligible for other frontline clinical trials of AML therapy. Prior therapy with hydroxyurea, hematopoietic growth factors, azacytidine, ATRA, or total dose of cytarabine up to 2g is allowed. Patients with history of MDS transformed to AML are eligible regardless of their prior therapy for MDS provided this will be their first induction therapy for AML.

9. Age >/= 18 years who are unsuitable for standard induction therapy are eligible after discussion with PI 10. Patients must have one of the following:

* Creatinine >/= 2 mg/dL
* Total bilirubin >/= 2 mg/dL
* ECOG Performance Status equal to 3 or 4
* Is ineligible for participation in a protocol of higher priority 11. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.

  12. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient is required prior to their enrollment on the protocol.

  13. Prior therapy with decitabine will be allowed unless the patient experienced progression to AML while being treated with decitabine.

Exclusion Criteria:

5. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.

6. Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, unless these illnesses are judged to be related to the underlying leukemia.

7. Patient with documented hypersensitivity to any of the components of the chemotherapy program.

8. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.

Cohort 3

Inclusion Criteria:

1. Patients with relapsed and or refractory AML who have received at least one prior therapy for their AML.
2. Age >/= 18 years.
3. Adequate organ function as defined below:

   * liver function (bilirubin < 2mg/dL, AST and/or ALT <3 x ULN)
   * kidney function (creatinine < 1.5 x ULN ).
4. ECOG performance status of ≤ 2.
5. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
6. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient is required prior to their enrollment on the protocol.
7. Prior therapy with venetoclax will be allowed.

   Exclusion Criteria
8. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
9. Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Patient with documented hypersensitivity to any of the components of the chemotherapy program.

Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-02-07 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Day 21
  Disease-free survival (DFS) defined as the time interval from treatment start until clinically significant disease progression or death, whichever occurred first. Participants followed for survival every 6 to 12 months after completion of active treatment. Study continuously monitored for primary endpoint, DFS using the method of Thall, Wooten, and Tannir.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kadia TM, Cortes J, Ravandi F, Jabbour E, Konopleva M, Benton CB, Burger J, Sasaki K, Borthakur G, DiNardo CD, Pemmaraju N, Daver N, Ferrajoli A, Wang X, Patel K, Jorgensen JL, Wang S, O'Brien S, Pierce S, Tuttle C, Estrov Z, Verstovsek S, Garcia-Manero G, Kantarjian H. Cladribine and low-dose cytarabine alternating with decitabine as front-line therapy for elderly patients with acute myeloid leukaemia: a phase 2 single-arm trial. Lancet Haematol. 2018 Sep;5(9):e411-e421. doi: 10.1016/S2352-3026(18)30132-7. Epub 2018 Aug 13. PMID 30115541
- See also: MD Anderson Cancer Center — http://www.mdanderson.org